CLINICAL TRIAL: NCT06608459
Title: Open-Label, Single Arm Study of PEX010-Assisted Therapy for Opioid Use Disorder (OUD): a Feasibility Study
Brief Title: PEX010-Assisted Therapy for Opioid Use Disorder (OUD): a Feasibility Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Filament Health Corp. (Industry)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PATOUD_F
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult participants with confirmed OUD (Experimental)
  Interventions: Drug: PEX010-Assisted Therapy

INTERVENTIONS:
Drug: PEX010-Assisted Therapy — The investigational medicinal product PEX010 is a capsule for oral administration that contains the drug substance PYEX.
  Other Names: PEX010

SUMMARY:
The goal of this clinical trial is to learn if it is feasible to use PEX010 for the treatment of opioid use disorder in adults. The study will also assess the safety of PEX010. The main questions it aims to answer are:

Can we successfully recruit participants, provide the drug and retain participants for the duration of the study?

What medical problems do participants experience when taking PEX010?

Participants will:

Take PEX010 twice during the study Engage in cognitive behavioural therapy Visit the clinic once or twice per week for study intervention and followup visits

DETAILED DESCRIPTION:
In this open-label study participants will receive PEX010, standardized to contain 25mg or 35 mg psilocybin, in conjunction with therapy. An open-label design was chosen given the novelty of this approach in treating OUD and high risk associated with opioid use.

Following screening and baseline visits, participants will receive 3 preparation sessions with psychotherapy, 2 PEX010 sessions, 2 integration sessions with psychotherapy, and 3 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed moderate to severe opioid use disorder as determined by the Mini-International Neuropsychiatric Interview (MINI), and the study physician assessment
* Have stable housing
* Have a local support person (close friend or family member) that is available to accompany them home
* If they are a person able to become pregnant (PABP):
* Be of non-childbearing potential, defined as (i) self-reported postmenopausal status (12 months of spontaneous amenorrhea and 45 years of age or older); or (ii) documented surgical sterilization (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy); or
* Have a negative pregnancy test at screening and prior to each PEX010 session, and must agree to use adequate contraception through 10 days after the last PEX010 session. Adequate contraception methods include intrauterine devices, oral hormones plus barrier contraception, abstinence, injectable or implanted hormonal methods, or vasectomized/non-sperm carrying sole partner. Barrier methods alone are not considered effective methods of contraception.
* Be willing to refrain from caffeine for minimum 12 hours, cannabis and alcohol for minimum 24 hours and all other drugs for at least 5 days prior to PEX010 administration such that there are no clinical signs of intoxication or withdrawal
* Be able and willing to follow study procedure
* Be able to understand, communicate and speak English
* Complete the Columbia Suicide Severity Rating Scale (CSSRS)
* Results from safety laboratory tests (CBC, AST and ALT, TSH, HbA1c) are within normal limits.

Exclusion Criteria:

* Are experiencing or at risk for significant withdrawal
* Have a history of overdose with opioids within the last 10 years
* Have any medical condition that would be contraindicated, including previously diagnosed conditions:
* seizure disorder or history of seizures;
* a history of significantly impaired hepatic function;
* a history of unstable or uncontrolled cardiovascular disease (coronary artery disease, heart failure, clinically significant ECG abnormality);
* uncontrolled hypertension, resting blood pressure greater than 140/90 mmHg;
* baseline prolongation of QTc interval greater than 450 msec in both males and females;
* a history of major central nervous system disease (history of cerebrovascular accident, masses, aneurysm);
* a history of uncontrolled obstructive airway disease or significant respiratory compromise;
* a history of uncontrolled thyroid disease;
* a history of uncontrolled insulin dependent diabetes that may preclude safe participation in the study;
* a history of narrow-angle glaucoma;
* gastrointestinal conditions which may affect psilocybin absorption (i.e. stenosing peptic ulcer, pyloroduodenal obstruction);
* a history of active obstructive urological conditions (i.e. symptomatic prostatic hypertrophy, bladder-neck obstruction) that may preclude safe participation in the study.
* Have any mental health disorder that would be contraindicated, including previously diagnosed or suspected mania/hypomania or psychosis as determined by the Modified MINI 7.0.1
* Have a first- or second-degree relative with psychotic or bipolar disorder
* Have a personality disorder deemed to be high risk (antisocial, borderline, narcissistic) assessed via the SCID-5-PD.
* Have a history of suicide attempt within the last 10 years or a suicidal ideation in the last year
* Have used any illicit stimulants or more than 3 drinks per week of alcohol in past 30 days
* Have used classic psychedelic drugs (e.g. psilocybin, LSD, DMT, ayahuasca, or mescaline) in the last 12 months or more than 25 times in lifetime, based on self-report
* Are currently taking medications with known interactions with psilocybin (e.g., antidepressants, antipsychotics)
* Are pregnant, breastfeeding, or they are a PABP and not practicing an adequate form of birth control
* Any other finding(s) based on the screening process that the investigator determines makes the candidate unsuitable for the study
* Results from safety laboratory tests (CBC, AST and ALT, TSH, HbA1c) are not within normal limits

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of AEs and SAEs | 8 weeks
  Total number of adverse events (AEs) and serious adverse events (SAEs) reported during the 8-week study period.

SECONDARY OUTCOMES:
Treatment retention | 8 weeks
  Percentage and number of participants who complete follow-up assessments.

IPD SHARING:
Plan to Share IPD: Undecided